CLINICAL TRIAL: NCT06582238
Title: Knowledge, Attitude and Practice for Management of Dentine Hypersensitivity Among Egyptian and Nigerian Dentists: A Cross-Sectional Comparative Study
Brief Title: Dentine Hypersensitivity Management KAP Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Muhammad Modu (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor
Other Study IDs: HypersensitivityCross
Record Dates: First submitted 2024-08-23; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Dentin Sensitivity
MeSH Terms: conditions — Dentin Sensitivity | interventions — Dentists

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Egyptian Dentists: Dentists (at various levels of education and years of practice) practicing in Egypt
  Interventions: Other: Dentists in Clinical Practice
- Nigerian Dentists: Dentists (at various levels of education and years of practice) practicing in Nigeria
  Interventions: Other: Dentists in Clinical Practice

INTERVENTIONS:
Other: Dentists in Clinical Practice — Experience in managing Dentine Hypersensitivity

SUMMARY:
The study aims to assess and compare the knowledge, attitudes, and practices of Egyptian and Nigerian dentists on etiology, diagnosis, and management of DH. Also to identify if level of education, culture and environment have influence in the diagnosis and management of DH.

DETAILED DESCRIPTION:
Diagnosis of dentin hypersensitivity is a challenge faced by dentists with different educational levels and the condition might be overlooked and not properly managed leading to persistent pain and poor quality of life for patients. Till the now, literature lacks rigorous guidelines for systematic diagnosis, prevention, categorization of severity and management of dentin hypersensitivity.

This study intends to spot the light on the current approaches adopted by dentists in Egypt and Nigeria towards diagnosis and management of Dentine Hypersensitivity. It also intends to compare the findings and identify the influence of geographic location, different educational levels, and degree of dental education in the management of Dentine Hypersensitivity

ELIGIBILITY:
Inclusion Criteria:

* Must be a Dentist
* Must be in clinical practice
* Must be practicing in Egypt or Nigeria
* Willingly CHOOSE to participate in the study

Exclusion Criteria:

* Dentists that choose NOT to participate in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Levels of Education
  * Consultant/Fellow/Professor
  * Specialist/Senior Lecturer
  * Resident/Registrar/Post Graduate Student
  * BDS
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-21 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 6 months
  % of Dentists with adequate knowledge of appropriate etiology diagnosis and management of DH among practicing dentists in Egypt and Nigeria using a validated questionnaire with options of various etiologies, diagnosis and management options. the subject chooses yes, no or i don't know.

SECONDARY OUTCOMES:
Comparison | 6 months
  Comparison of Knowledge and management practices of dentists in Egypt and Nigeria in the management of dentine sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-07-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT06582238/Prot_ICF_000.pdf